CLINICAL TRIAL: NCT00705744
Title: Dermatological Evaluation of the Photo Irritation and Photo Sensitivity Potential for Dermacyd Femina.
Brief Title: Dermacyd Femina (Lactic Acid) - Photo Dermatological Evaluation of the Irritation and Sensitivity Potential.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_03982
Record Dates: First submitted 2008-06-25; First posted 2008-06-26 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental)
  Interventions: Drug: Lactic acid (Dermacyd Femina)

INTERVENTIONS:
Drug: Lactic acid (Dermacyd Femina)

SUMMARY:
To prove the absence of photo irritation and photo sensitivity potential of the product Dermacyd Femina.

ELIGIBILITY:
Inclusion Criteria:

* Phototype Skin II and III;
* Integral skin test in the region;

Exclusion Criteria:

* Lactation or gestation;
* Use of Anti-inflammatory and/or immuno-suppression drugs 15 days before the selection;
* Diseases which can cause immunity decrease, such as HIV, diabetes;
* Use of drug photosensitizer;
* History of sensitivity or irritation for topic products;
* Active cutaneous disease which can change the study results;
* History or photodermatosis active;
* Family or personal antecedent of cutaneous photoinduced neoplasias;
* Presence of a precursor lesion of cutaneous neoplasia, such as nevus melanocyte and keratoses actinium;
* Intense solar exposure in the study area;
* Use of new drugs or cosmetics during the study;

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-04; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The photo irritation test and the photosensitivity will be measured using UVA irradiation and evaluated according International Contact Dermatitis Research Group (ICDRG) scale | 5 weeks
The sensibility will be evaluated according to the skin type. | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, MD, Study Director — Sanofi
Locations (1):
- Sanofi-aventis, São Paulo, São Paulo, Brazil